CLINICAL TRIAL: NCT03286400
Title: Observational Registry Characterizing the Performance and Feature Use of the GORE® TAG® Conformable Thoracic Stent Graft Featuring ACTIVE CONTROL System
Brief Title: Observational Registry Characterizing the CTAG Device With ACTIVE CONTROL
Acronym: SURPASS
Status: Completed | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: TAG 15-03
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Results first posted 2020-11-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Thoracic Diseases
Keywords: CTAG; TEVAR
MeSH Terms: conditions — Thoracic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CTAG Device with ACTIVE CONTROL: All consecutive patients meeting protocol selection criteria, consented, with an intention to be treated with CTAG Device with ACTIVE CONTROL.
  Interventions: Device: CTAG Device with ACTIVE CONTROL

INTERVENTIONS:
Device: CTAG Device with ACTIVE CONTROL — Intent to treat with the CTAG Device with ACTIVE CONTROL in the treatment of aortic diseases as part of routine clinical practice.

SUMMARY:
Collect real-world clinical and device-specific outcomes of the GORE® TAG® Conformable Thoracic Stent Graft featuring ACTIVE CONTROL System (CTAG Device with ACTIVE CONTROL) in the treatment of aortic disease as part of routine clinical practice.

DETAILED DESCRIPTION:
This is an observational, prospective, single-arm, post-market registry designed to collect real-world clinical and device specific outcomes of the GORE® TAG® Conformable Thoracic Stent Graft featuring ACTIVE CONTROL System (CTAG Device with ACTIVE CONTROL) in the treatment of aortic disease as part of routine clinical practice. A maximum of 20 clinical investigative sites in Europe will participate and up to 125 patients will be enrolled in this registry. All consecutive patients meeting protocol selection criteria, consented, with an intention to be treated with the CTAG Device with ACTIVE CONTROL will be included and followed through one year per institutional standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Signed informed consent form
3. Willingness, in the opinion of the investigator, to adhere to standard of care follow-up requirements
4. Surgical indication for TEVAR based on investigator's best medical judgment
5. Intent to treat with CTAG Device with ACTIVE CONTROL.

Exclusion Criteria:

1. Paraplegia or paraparesis at initial presentation
2. Participation in concurrent research study or registry which may confound registry results, unless approved by Sponsor
3. Prior implantation of a thoracic stent graft
4. Pregnant or breast-feeding female at time of informed consent signature
5. Life expectancy < 1 year due to comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients presenting with an indication for endovascular repair of the thoracic aorta are eligible for screening for participation in the registry. Only patients who meet all inclusion and no exclusion criteria, and who consent to participate will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Torsello, MD, PhD, Principal Investigator — St Franziskus Hospital GmbH
Locations (20):
- France (2):
  - University Hospital Angers, Angers
  - CHU Strasbourg, Strasbourg
- Germany (4):
  - University Hospital Köln, Cologne
  - University of Heidelberg, Heidelberg
  - St. Franziskus Hospital GmbH, Münster
  - University Hospital Regensburg, Regensburg
- Italy (3):
  - Hospital Civili Brescia, Brescia
  - Ospedali dei Colli - Monaldi, Napoli
  - Azienda Ospedaliers San Camilla Forlanni, Roma
- Netherlands (3):
  - University Hospital Amsterdam, Amsterdam
  - St Antonius Hospital, Nieuwegein
  - Erasmus Medical Center, Rotterdam
- Spain (3):
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Clínico Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (2):
  - Orebro University Hospital, Örebro
  - Uppsala University, Uppsala
- United Kingdom (3):
  - Leeds General Infirmary, Leeds
  - St George's Vascular Institute, London
  - St Thomas' London / Guy's Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Torsello GF, Argyriou A, Stavroulakis K, Bosiers MJ, Austermann M, Torsello GB; SURPASS Registry Collaborators. One-Year Results From the SURPASS Observational Registry of the CTAG Stent-Graft With the Active Control System. J Endovasc Ther. 2020 Jun;27(3):421-427. doi: 10.1177/1526602820913007. Epub 2020 Mar 20. PMID 32193990

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CTAG Device With ACTIVE CONTROL
Started | 127
Completed | 102
Not Completed | 25
Not completed — Death | 10
Not completed — Lost to Follow-up | 10
Not completed — Physician Decision | 1
Not completed — Scheduling difficulty | 4

BASELINE CHARACTERISTICS:
Arm/Group | CTAG Device With ACTIVE CONTROL
Number analyzed (Participants) | 127
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.1 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 92
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 33
  Sweden | 9
  Italy | 24
  United Kingdom | 5
  France | 7
  Germany | 39
  Spain | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Procedural Technical Success
Description: Successful access to the arterial system, successful deployment at the intended location, patent endoluminal graft, absence of surgical conversion
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | CTAG Device With ACTIVE CONTROL
Number analyzed (Participants) | 127
Participants | 123

2. Primary Outcome: Number of Subjects With Treatment Success at 30 Day Visit
Description: Technical Success and Freedom from: Type I or III endoleak, rupture of lesion in treated segment, stent graft occlusion, stent graft migration
Time Frame: One month
Population: Includes all subjects with treatment failure within 30 days as well as subjects with at least 15 days of follow-up. Subjects without a treatment failure within 30 days and with less than 15 days of follow-up were not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CTAG Device With ACTIVE CONTROL
Number analyzed (Participants) | 125
Participants | 115

3. Secondary Outcome: Number of Subjects With Freedom From Major Adverse Events at 30 Days
Description: Freedom from: Lesion-related mortality, permanent paraplegia or paraparesis, disabling stroke, life-threatening myocardial infarction, new onset of renal failure, respiratory failure, life-threatening bowel ischemia, serious tissue ischemia, major blood loss
Time Frame: 30 Days
Population: Includes all subjects with a Major Adverse Event within 30 days as well as subjects with at least 15 days of follow-up. Subjects without a Major Adverse Event within 30 days and with less than 15 days of follow-up were not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CTAG Device With ACTIVE CONTROL
Number analyzed (Participants) | 116
Participants | 105

4. Secondary Outcome: Number of Subjects With Freedom From Major Adverse Events at 12 Months
Description: as for outcome 3
Time Frame: 12 Months
Population: Includes all subjects with a Major Adverse Event within 12 months as well as subjects with at least 275 days of follow-up. Subjects without a Major Adverse Event within 12 months and with less than 275 days of follow-up were not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CTAG Device With ACTIVE CONTROL
Number analyzed (Participants) | 102
Participants | 90

5. Secondary Outcome: Number of Subjects With Treatment Success at 12 Month Visit
Description: Technical Success and Freedom from: Type I or III endoleak, rupture of lesion within treated segment, stent graft occlusion, stent graft migration
Time Frame: One year
Population: Includes all subjects with treatment failure within 12 months as well as subjects with at least 275 days of follow-up. Subjects without a treatment failure within 12 months and with less than 275 days of follow-up were not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CTAG Device With ACTIVE CONTROL
Number analyzed (Participants) | 111
Participants | 97

6. Secondary Outcome: Probability of Freedom From Serious Adverse Events, Other Than Major Adverse Events
Description: Freedom from incidence of Serious Adverse Events, other than Major Adverse Events, throughout the Registry Duration. Estimates determined from Kaplan-Meier analysis.
Time Frame: Days 30, 365, and 455
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | CTAG Device With ACTIVE CONTROL
Number analyzed (Participants) | 127
Probability
  30 Days | 0.826 [0.748 to 0.882]
  365 Days | 0.699 [0.609 to 0.772]
  455 Days | 0.628 [0.487 to 0.740]

7. Secondary Outcome: Change in Maximum Aortic Diameter Among Aneurysm/Isolated Lesion
Description: One year change from first post-implant CT scan in maximum aortic diameter
Time Frame: One year
Population: Includes all non-dissection subjects who have both post-procedure and 12-month measurements.
Measure: Count of Participants; unit: Participants
Arm/Group | CTAG Device With ACTIVE CONTROL
Number analyzed (Participants) | 47
Participants
  >= 5mm Decrease | 20
  No Change | 22
  >= 5mm Increase | 5

8. Secondary Outcome: Change in Maximum False Lumen Diameter Among Dissection
Description: One year change from first post-implant CT scan in maximum false lumen diameter
Time Frame: One year
Population: Includes all dissection subjects who have both post-procedure and 12-month measurements.
Measure: Count of Participants; unit: Participants
Arm/Group | CTAG Device With ACTIVE CONTROL
Number analyzed (Participants) | 26
Participants
  >= 5mm Decrease | 15
  No Change | 10
  >= 5mm Increase | 1

9. Secondary Outcome: Change in Minimum True Lumen Diameter Among Dissection
Description: One year change from first post-implant CT scan in minimum true lumen diameter
Time Frame: One year
Population: Includes all dissection subjects who have both post-procedure and 12-month measurements.
Measure: Count of Participants; unit: Participants
Arm/Group | CTAG Device With ACTIVE CONTROL
Number analyzed (Participants) | 26
Participants
  >= 5mm Decrease | 5
  No Change | 11
  >= 5mm Increase | 10

10. Secondary Outcome: Change in Maximum Aortic Diameter Among Dissection
Description: One year change from first post-implant CT scan in maximum aortic diameter
Time Frame: One year
Population: Includes all dissection subjects who have both post-procedure and 12-month measurements.
Measure: Count of Participants; unit: Participants
Arm/Group | CTAG Device With ACTIVE CONTROL
Number analyzed (Participants) | 26
Participants
  >= 5mm Decrease | 14
  No Change | 10
  >= 5mm Increase | 2

ADVERSE EVENTS:
Time Frame: 455 days
Arm/Group | CTAG Device With ACTIVE CONTROL
All-Cause Mortality (participants affected / at risk) | 10/127
Serious Adverse Events (participants affected / at risk) | 45/127
Other Adverse Events (participants affected / at risk) | 0/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CTAG Device With ACTIVE CONTROL (N=127)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Aorto-oesophageal fistula (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Stent-graft endoleak (General disorders) | 9 (10)
Vascular stent occlusion (General disorders) | 1 (1)
Infective aneurysm (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Vascular device infection (Infections and infestations) | 1 (1)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Vascular graft haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Vascular procedure complication (Injury, poisoning and procedural complications) | 2 (2)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1)
Pancreatogenous diabetes (Metabolism and nutrition disorders) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Paraplegia (Nervous system disorders) | 2 (2)
Spinal cord ischaemia (Nervous system disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Diaphragmatic disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Aortic aneurysm (Vascular disorders) | 3 (3)
Aortic dissection (Vascular disorders) | 3 (3)
Aortic rupture (Vascular disorders) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT03286400/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT03286400/SAP_001.pdf